CLINICAL TRIAL: NCT03606135
Title: Etiology and Incidence Assessment of Radiographically-confirmed Community Acquired Pneumonia (CAP) in Adults ≥ 18 Years (OSPIS)
Brief Title: Etiology and Incidence Assessment of Radiographically-confirmed Community Acquired Pneumonia (CAP)
Acronym: OSPIS
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/220
Record Dates: First submitted 2018-07-09; First posted 2018-07-30 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia
Keywords: Pneumonia; Streptococcus pneumoniae; Incidence; Ethiology; Serotype
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal samples (flocked swab), oral samples (flocked swab), urine and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Pneumonia Group: Subjects with chest images (x-ray or CT scan) indicating pneumonia.
  Interventions: Other: The Pneumonia Group
- The Control Group: Healthy subjects
  Interventions: Other: The Control Group

INTERVENTIONS:
Other: The Pneumonia Group
  Groups: The Pneumonia Group
Other: The Control Group
  Groups: The Control Group

SUMMARY:
This is an epidemiological study to investigate the etiology of radiographically-confirmed community-acquired pneumonia (CAP) in adults aged ≥18 years. The main objective is to determine the proportion of which cases that is due to Streptococcus pneumoniae and the corresponding incidence and serotype distribution. The study will utilize a serotype-specific urinary antigen detection (UAD) assay.

ELIGIBILITY:
The Pneumonia Group

Inclusion Criteria:

* Age ≥ 18 years.
* Present to a study healthcare facility where treating physician clinically suspects CAP with the presence of two or more of the following signs and symptoms: Fever, Hypothermia, Chills or rigors, Pleuritic chest pain, Cough, Sputum production, Dyspnea, Tachypnea, Malaise, Abnormal auscultatory findings suggestive of pneumonia.
* Has radiographic finding that is consistent with pneumonia.
* Able and willing to provide urine sample.
* Signed and dated informed consent

Exclusion Criteria:

* Transferred to a study healthcare facility after already being hospitalized for 48 hours or more at any other in-patient facility.
* Hospital acquired pneumonia.
* Subjects who are investigational staff members and their family members, and site staff members otherwise supervised by the investigator.
* Previous enrollment in this study within the previous 30 days.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.

The Control Group

Inclusion Criteria:

* Signed and dated informed consent.
* Age ≥ 18 years.
* Able and willing to provide urine sample.

Exclusion Criteria:

* Subjects who are investigational staff members or relatives of those staff member or subjects who are Pfizer employees directly involved in the conduct of the study.
* Subjects with suspicion of CAP or any other respiratory infectious disease, as well as evidence of or documented concomitant infectious disease.
* Subjects residing in any long-term care facilities.
* Subjects with known bronchial obstruction or history of post-obstructive pneumonia. Chronic obstructive pulmonary disease (COPD) is permissible, provided there has no been an exacerbation with 3 months prior to enrollment.
* Subjects with primary lung cancer or another malignancy metastatic to the lungs.
* Subjects with fever.
* Subjects with significant immunosuppressive disease such as AIDS, leukemia, etc.
* Subjects with either pneumococcal conjugate vaccine (PCV) and/or pneumococcal polysaccharide vaccine (PPV) administration within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Pneumonia Group: Adults ≥ 18 years of age who present to the emergency room with signs and symptoms of CAP and have radiographic evidence of pneumonia, as read by the clinical radiologist on duty will be identified and enrolled. As this is an active, prospective surveillance study, all eligible subjects should be screened for enrolment, including whose who are admitted during nights.
  The Control Group: Subjects will be sceened by the nurse at the orthopedic section of the emergency unit, since these patients are unlikely to have respiratory tract infections. Subjects will be chosen randomly and evenly over the whole duration of the study to get a representative control group.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-09-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion S.pneumoniae serotypes included in PCV13 (Pneumococcal conjugate vaccine) among adults ≥18 years of age presenting with radiographically-confirmed CAP. | 10 days
  The overall proportion of subjects with clinically and radiographically-confirmed CAP who have PCV13 S.pneumoniae detected by either UAD assay and/or culture.

SECONDARY OUTCOMES:
The S.pneumoniae serotype distribution form UAD and culture isolates. | 10 days
  The full distribution of all S.pneumoniae serotypes among patients with CAP.
The incidence rate of CAP and subjects with S.pneumoniae positive radiologically confirmed CAP (SP+CAP) | 10 days
  The incidence rate of CAP and SP+CAP
The differences in detection of S.pneumoniae by culture, BinaxNOW® and the UAD assay | 10 days
  The overall proportion of SP+CAP subjects with S.pneumoniae identified by culture, BinaxNOW®, and/or either UAD assay.
The proportion of subjects with CAP and with SP+CAP who present with underlying at-risk and high-risk medical conditions | 10 days
  The proportion of subjects with CAP and SP+CAP who present with underlying at-risk and high-risk medical conditions.
Antibiotic resistance rates among isolates of S.pneumoniae | 10 days
  Antibiotic resistance rates among isolates of S.pneumoniae.
Validation of the UAD assay in CAP patients and compare with controls | 10 days
  To validate the UAD assay in CAP patients and compare results with the control group.

OTHER OUTCOMES:
Distribution of different microbial findings in subjects with CAP including the proportion of co-infection and correlate with severity of disease | 10 days
  To define the distribution of different microbial findings in subjects with CAP and estimate viral and bacterial load using semi-quantitive PCR and correlate it with severity of disease and calculate the proportion of subjects with co-infection.
Difference in sensitivity in detection of bacterial agents, comparing sputum and nasopharyngeal sampling and comparing bacterial culture with PCR | 10 days
  To define the difference in sensitivity in detection of bacterial agents, comparing sputum and nasopharyngeal sampling and comparing bacterial culture with PCR (Polymerase Chain Reaction).
Distribution of nasopharyngeal microbial findings in subjects with CAP in comparison to an asymptomatic control group | 10 days
  To determine differences in nasopharyngeal microbial findings in subjects with CAP and an asymptomatic control group.
The microbiome in the respiratory tract in subjects initially diagnosed with CAP and after 3 months. The control group will be included. | 3 months
  To determine the microbiome in the respiratory tract in subjects diagnosed with CAP and compare those microbiomes 3 months later. CAP subjects will be compared with the control group.
Antibiotic resistance rate of bacterial isolates | 10 days
  To estimate antibiotic resistance rates among bacterial isolates, other than S.pneumoniae.
Correlation of antibiotic regimen, clinical outcome and readmission | 3 months
  To calculate the correlation of antibiotic regimen, ICU, length-of-stay (LOS) and clinical outcome including mortality after 90 days in addition to readmission rate.
Etiology and and outcome in patients with CAP and correlate it to the Charlson Comorbidity Index, CRB-65, and Pneumonia Severity Index | 3 months
  Etiology and and outcome in patients with CAP and correlate it to the Charlson Comorbidity Index, CRB-65 (Confusion-Rate-Blood pressure, ≥65 years) and Pneumonia Severity Index
Correlation between treatment with protein pump inhibitors and CAP | 10 days
  To observe any correlation between CAP and treatment with protein pump inhibitors.
Correlation of the levels of vitamin D and severity of CAP | 10 days
  To correlate levels of vitamin D to severity of CAP
New cognitive impairment at follow-up | 3 months
  To determine which factors of MoCA (Montreal Cognitive Assessment) are associated with long-term cognitive impairment after hospitalization with pneumonia.
Newly acquired functional disability of performing physical activities at follow-up | 3 months
  To determine which factors of P-ADL (Physical Activities of Daily Living) are associated with functional decline after pneumonia.
Newly acquired functional disability of performing instrumental activities at follow-up | 3 months
  To determine which factors of I-ADL (Instrumental Activities of Daily Living) are associated with functional decline after pneumonia.
Decline in quality of life from enrolment to follow-up | 3 months
  To determine which factors of EQ-5D (European Quality of life - 5 Dimensions) are associated with declining quality of life after pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Ahl, MD, PhD, Principal Investigator — Department of Infectious Diseases
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansen K, Yamba Yamba L, Wasserstrom L, Runow E, Goransson T, Nilsson A, Ahl J, Riesbeck K. Exploring the microbial landscape: uncovering the pathogens associated with community-acquired pneumonia in hospitalized patients. Front Public Health. 2023 Dec 13;11:1258981. doi: 10.3389/fpubh.2023.1258981. eCollection 2023. PMID 38152664